CLINICAL TRIAL: NCT02493361
Title: An Open-label, Phase II, Multicenter Study of Enhancing Pembrolizumab Responses in Melanoma Through Intratumoral pIL-12 Electroporation
Brief Title: Trial of pIL-12/MK-3475 in Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: OncoSec Medical Incorporated (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Katy Tsai, Clinical Assistant Professor, University of California, San Francisco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15852; NCI-2015-01300 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2015-07-06; First posted 2015-07-09 (Estimated); Results first posted 2019-08-21 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2020-12

CONDITIONS: Melanoma
Keywords: Pembrolizumab; Intratumoral pIL-12 Electroporation; Tumor-infiltrating lymphocyte melanoma
MeSH Terms: conditions — Melanoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Pembrolizumab: 200 mg IV, Day 1 of each cycle pIL-12: 1/4 tumor volume at concentration of 0.5 mg/mL intratumoral, Days 1, 5, and 8 of each odd cycle
  Interventions: Drug: Pembrolizumab; Drug: pIL-12

INTERVENTIONS:
Drug: Pembrolizumab
Drug: pIL-12

SUMMARY:
This is a multicenter, Phase II, open-label, 42-patient single-arm trial of intratumoral pIL-12 electroporation (EP) in combination with pembrolizumab in patients with melanoma. Patients will be evaluated in 2 parts. Part A patients will be selected using a flow cytometric assay that quantifies intratumoral PD-1hiCD8+CTLA4+ "exhausted" lymphocytes in the tumor. Part B will enroll patients who have or are failing pembrolizumab at least 12 weeks after starting Programmed cell death protein 1 (PD-1) antibody alone or in combination, or, who have been selected using a flow cytometric assay that quantifies intratumoral PD-1hiCD8+CTLA4+ "exhausted" lymphocytes in the tumor.

DETAILED DESCRIPTION:
Closed to enrollment earlier than expected due to high response rate in order to advance to phase 2b in proven PD-1-refractory patients. A total of 24 patients were consented instead of the planned enrollment of 42 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histological or cytological diagnosis of melanoma with progressive locally advanced or metastatic disease that is not amenable to definitive local therapy with curative intent.
* At least one measurable tumor accessible for intratumoral injection and EP on investigator's assessment.
* Patients may have had prior chemotherapy or immunotherapy or radiation therapy. All prior therapies must be stopped 4 weeks prior to first dose of study treatment, with the exception of patients who have received ipilimumab, which must be stopped 6 weeks prior to first dose of study treatment. Patients are prohibited from receiving live vaccines within 30 days prior to first dose of study treatment.
* Age >= 18 years
* Part A: Patient has agreed to two newly obtained tumor biopsies and as required re-biopsies (that can be biopsied on investigator's assessment) and to providing the acquired tissue for biomarker analysis. Analysis of one of the fresh biopsy samples for PD-1hiCD8+CTLA4hi in the CD8+CD45+ gate based on flow cytometry will be done. A second fresh biopsy sample is required for further biomarker analysis and confirmation at a later date of low PD-L1 expression using an Immunohistochemistry (IHC) assay for PD-L1 expression. A valid flow cytometry result is not required for study participation, but repeated biopsy for reanalysis is strongly recommended for patient with insufficient tumor-infiltrating lymphocytes (TIL) in the first tissue sample. Or:
* Part B: Anti-PD-1 non-responders are defined as those showing disease progression according to RECIST v1.1 after at least 12 weeks of therapy with a PD-1 antibody either alone or in combination with approved checkpoint inhibitor or targeted therapies according to their label. There is no serological requirement.
* Life expectancy of at least 6 months.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Adequate organ function within 4 weeks of administration of study therapy:

  1. Lactate dehydrogenase (LDH): <4 x upper limit of normal (ULN)
  2. Adequate hematological function:

     1. Absolute neutrophil count (ANC): >=1,500/μL
     2. Platelets: >=100,000/μL
     3. Hemoglobin: >= 9 g/dL
  3. Adequate hepatic function:

     1. Serum total bilirubin: ≤1.5 x ULN OR Direct bilirubin <= ULN for patients with total bilirubin levels >1.5 ULN
     2. aspartate aminotransferase (AST) / serum glutamic-oxaloacetic transaminase (SGOT) and alanine aminotransferase (ALT) / serum glutamic-pyruvic transaminase (SGPT): <=2.5 x ULN OR ≤5 x ULN for patients with liver metastases
  4. Adequate renal function:

     1. Serum creatinine: ≤1.5 x ULN
  5. Coagulation:

     1. International normalized ration (INR) or Prothrombin Time (PT): ≤1.5 x ULN (Only if not using anticoagulants. If patient is receiving anticoagulants, then value must be within therapeutic range for the condition that patient is being treated for).
     2. Activated partial thromboplastin time (aPTT): <=1.5 x ULN (Only if not using anticoagulants. If patient is receiving anticoagulants, then value must be within therapeutic range for the condition that patient is being treated for).
* Female patient of childbearing potential has a negative serum or urine pregnancy test within 14 days prior to administration of study therapy.
* The effects of pIL-12 EP and pembrolizumab on the developing human fetus are unknown. For this reason women of child-bearing potential (not free from menses for >2 years, post hysterectomy/oophorectomy, or surgically sterilized) must agree to use two methods of contraception, or abstain from heterosexual activity, during participation in study, from the time of consent through 120 days after the last dose of study therapy. The two methods must include at least one "barrier method". Barrier methods are diaphragms, cervical caps, cervical shields, male condoms, and female condoms. The second method of contraception may be another barrier method, a copper containing intrauterine device (IUD), spermicidal foams, sponges and films, or hormone-based contraception (for example, hormone pills, hormone rings, hormone patches, hormone-releasing IUDs, or Depo Provera). Men with partners who are capable of getting pregnant must agree to use one of the barrier methods of contraception listed above during participation in the study, starting with the first dose of study drug through 120 days after the last dose of study therapy. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Ability to understand a written informed consent document, and the willingness to sign and date it.

Exclusion Criteria:

* Patient is currently participating or has participated in a study of an investigational agent or using an investigational device within 4 weeks of administration of study therapy.
* Patient is expected to require any other form of antineoplastic therapy while on study; including systemic chemotherapy, biological therapy, immunotherapy not specified in this protocol.
* Patient has uveal melanoma.
* Patient has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided they are clinically stable without the use of systemic steroids for at least 8 weeks prior to study entry.
* Patient has risk factors for bowel obstruction or bowel perforation (examples include but not limited to a history of acute diverticulitis, intra-abdominal abscess, and abdominal carcinomatosis).
* Patient previously had a severe hypersensitivity reaction to treatment with another monoclonal antibody (mAb).
* Patient has a history of history of (non-infectious) pneumonitis or interstitial lung disease.
* Patient has active infection at time of study entry that require systemic antibiotics and/or with an oral temperature of >= 38.3 degrees Celsius (°C)(100.9 degrees Fahrenheit (°F)) within 5 days of first treatment.
* Patients with electronic pacemakers or defibrillators are excluded from this study, as the effect of electroporation on these devices is unknown. Patients with lower extremity lesions may be discussed with the medical monitor.
* Patient has an active autoimmune disease or a documented history of autoimmune disease or syndrome that requires systemic steroids or immunosuppressive agents. Patients with vitiligo or resolved childhood asthma/atopy would be exception to this rule. Patients that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Patients with hypothyroidism that is stable on hormone replacement will not be excluded from the study.
* Patient has a medical condition that requires chronic systemic steroid therapy or requires any other form of immunosuppressive medication. However, patients using physiologic replacement doses of hydrocortisone, or its equivalent, will be considered eligible for this study; up to 20 mg hydrocortisone (or 5 mg of prednisone) in the morning and 10 mg hydrocortisone (or 2.5 mg of prednisone) in the evening.
* Pregnant women are excluded from this study because the potential for teratogenic or abortifacient effects upon treatment with pIL-12 EP + pembrolizumab is unknown. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with pIL-12 EP + pembrolizumab breastfeeding should be discontinued if the mother is treated with pIL-12 EP + pembrolizumab.
* Patients with symptomatic ascites or pleural effusion. A patient who is clinically stable following treatment for these conditions is eligible.
* Patient is Hepatitis C Virus (HCV) Ab positive or HBSAg positive.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-08-17 (Actual); Primary Completion 2018-04-26 (Actual); Study Completion 2020-03-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katy Tsai, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - University of San Francisco, California, San Francisco, California
  - Huntsman Cancer Institute, University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jacobs L, Yshii L, Junius S, Geukens N, Liston A, Hollevoet K, Declerck P. Intratumoral DNA-based delivery of checkpoint-inhibiting antibodies and interleukin 12 triggers T cell infiltration and anti-tumor response. Cancer Gene Ther. 2022 Jul;29(7):984-992. doi: 10.1038/s41417-021-00403-8. Epub 2021 Nov 9. PMID 34754076

RESULTS

PARTICIPANT FLOW:
Groups:
- Pembrolizumab and Intratumoral pIL-12 Electroporation: Treatments of pembrolizumab and pIL-12 were given in three week cycles that repeated as long as there was benefit, for up to 24 months or until disease worsened. Some subjects had the option of continuing treatment beyond 24 months or after worsening of disease under limited circumstances.
  Pembrolizumab: 200 mg dose is given intravenously, Day 1 of each cycle. pIL-12: Given by injection into the tumor at 1/4 tumor volume at concentration of 0.5 mg/mL, Days 1, 5, and 8 of each odd numbered cycle.
Period: Overall Study
Arm/Group | Pembrolizumab and Intratumoral pIL-12 Electroporation
Started | 24
Week 24 Assessment | 21
Completed | 21
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab and Intratumoral pIL-12 Electroporation
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.5 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 21
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Objective Response Rate (ORR) Within 24 Weeks Using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Description: Best overall ORR within 24 weeks of first treatment with pIL-12 electroporation (EP) and pembrolizumab will be determined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT or MRI. The ORR is the proportion of participants with either a Complete Response (CR) defined as a disappearance of all target lesions determined by 2 separate scans conducted not < 4 weeks apart and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm (the sum may not be "0" if there are target nodes) and no appearance of new lesions or a Partial Response (PR) defined as a >=30% decrease in the sum of the longest diameter of target lesions with no appearance of new lesions. ORR = CR + PR.
Time Frame: Up to week 24
Measure: Number; unit: proportion of participants
Arm/Group | Pembrolizumab and Intratumoral pIL-12 Electroporation
Number analyzed (Participants) | 24
proportion of participants | 0.375

2. Secondary Outcome: Best Overall ORR Determined by Immune Related-Response Criteria (irRC)
Description: Best overall objective response rate is defined as the proportion of participants with a demonstrated complete or partial response according to irRC. In the irRC, an immune-related Complete Response (irCR) is the disappearance of all lesions, measured or unmeasured, and no new lesions; an immune-related Partial Response (irPR) is a 50% drop in tumour burden from baseline as defined by the irRC.
Time Frame: Up to 5 years
Measure: Number; unit: proportion of participants
Arm/Group | Pembrolizumab and Intratumoral pIL-12 Electroporation
Number analyzed (Participants) | 21
proportion of participants | .429

3. Secondary Outcome: Twenty-Four Week Landmark Progression Free Survival (PFS)
Description: Twenty-four week landmark PFS (PFS at 24) is defined as the percentage of patients, who have progressed at the 24 week time point (+ / - 2 days visit tolerance). Tumor response determinations were assessed by RECIST v1.1.
Time Frame: At 24 weeks after treatment initiation
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Pembrolizumab and Intratumoral pIL-12 Electroporation
Number analyzed (Participants) | 21
days | 170 [86 to 170]

4. Secondary Outcome: Number of Participants With Treatment-related Adverse Events
Description: The study will use the NCI Common Terminology Criteria for Adverse Events (CTCAE) v4.0 with an adverse or serious adverse event determination of possible, probable, or definite attribution. Analyses will be performed for all patients having received at least one dose of study drug.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab and Intratumoral pIL-12 Electroporation
Number analyzed (Participants) | 24
Participants | 2

5. Secondary Outcome: Median PFS
Description: PFS is defined as the duration between the date of treatment initiation to the first date of either disease progression where progression is assessed by RECIST v1.1, or death.
Time Frame: Up to 5 years
Measure: Median (Full Range); unit: days
Arm/Group | Pembrolizumab and Intratumoral pIL-12 Electroporation
Number analyzed (Participants) | 21
days | 253 [86 to 1659]

6. Secondary Outcome: Duration of Response (DOR) Estimate
Description: DOR is defined as the number of days from the initial documentation of an objective response (CR or PR) per RECIST v1.1 criteria to the final evaluation of that response (censored duration), or to documentation of progression using Kaplan-Meier (KM) estimates .
Time Frame: Up to 5 years
Measure: Number; unit: months
Arm/Group | Pembrolizumab and Intratumoral pIL-12 Electroporation
Number analyzed (Participants) | 9
months | NA — Of the 9 participants with an objective response (CR or PR), 0 patients progressed after achieving an objective response and therefore all of the durations were censored. As a result, the KM estimates are not calculable.

7. Secondary Outcome: Overall Survival (OS) Estimate
Description: OS is defined as the duration between the date of treatment initiation to the date of death, regardless of the cause of death using KM estimates.
Time Frame: Up to 5 years
Measure: Number; unit: days
Arm/Group | Pembrolizumab and Intratumoral pIL-12 Electroporation
Number analyzed (Participants) | 24
days | NA — The KM estimate could not be calculated given that 82% of the subjects were still alive at the time of the last follow-up and over 80% of the OS durations were censored.

ADVERSE EVENTS:
Time Frame: Up to 5 years
Arm/Group | Pembrolizumab and Intratumoral pIL-12 Electroporation
All-Cause Mortality (participants affected / at risk) | 4/24
Serious Adverse Events (participants affected / at risk) | 3/24
Other Adverse Events (participants affected / at risk) | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab and Intratumoral pIL-12 Electroporation (N=24)
Skin infection (Infections and infestations) | 1 (1) — Cellulitis
Myocardial infarction (Cardiac disorders) | 1 (1)
Hepatobiliary disorders - Other (Hepatobiliary disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab and Intratumoral pIL-12 Electroporation (N=24)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Alkaline phosphatase increased (Investigations) | 2 (2)
Creatinine increased (Investigations) | 3 (3)
Lactate dehydrogenase increased (Investigations) | 2 (2)
Thyroid stimulating hormone increased (Investigations) | 2 (2)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Bronchitis
Constipation (Gastrointestinal disorders) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Anorexia (Metabolism and nutrition disorders) | 3 (3) — Decreased appetite
Depression (Psychiatric disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Dizziness (Nervous system disorders) | 9 (9)
Fatigue (General disorders) | 17 (17)
Fall (General disorders) | 3 (3)
Headache (Nervous system disorders) | 5 (5)
Hypoesthesia (Nervous system disorders) | 3 (3)
Flu like symptoms (General disorders) | 2 (2)
Injection site pain (Injury, poisoning and procedural complications) | 3 (3)
Insomnia (Psychiatric disorders) | 2 (2)
Muscle spasm (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 8 (8)
Peripheral edema (General disorders) | 5 (5)
Procedural pain (Injury, poisoning and procedural complications) | 13 (13)
Pruritus (Skin and subcutaneous tissue disorders) | 8 (8)
Fever (General disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Rash pruritic (Skin and subcutaneous tissue disorders) | 7 (7)
Sinusitis (Infections and infestations) | 2 (2)
Tremor (Nervous system disorders) | 2 (2)
Blurred vision (Eye disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 2 (2)
Weight loss (Investigations) | 2 (2)
Hematocrit decreased (Blood and lymphatic system disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
Closed to enrollment earlier than expected due to high response rate in order to advance to phase 2b in proven PD1-refractory patients. A total of 24 patients were consented instead of the planned enrollment of 42 patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-06): https://cdn.clinicaltrials.gov/large-docs/61/NCT02493361/Prot_SAP_000.pdf